CLINICAL TRIAL: NCT03480685
Title: A Post-market, Multi-vessel Evaluation of the Imaging of Peripheral Arteries for Diagnostic Purposes Comparing Optical Coherence Tomography and Intravascular Ultrasound Imaging
Brief Title: Evaluation of Imaging of Peripheral Arteries by Optical Coherence Tomography and Intravascular Ultrasound Imaging
Acronym: SCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P0986
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IVUS Imaging vs. OCT Imaging (Other): A vessel segment will be imaged with intravascular ultrasound (IVUS). The same vessel segment will be imaged with optical coherence tomography (OCT).
  Interventions: Device: IVUS and OCT Imaging

INTERVENTIONS:
Device: IVUS and OCT Imaging — Use of an imaging catheter

SUMMARY:
A non inferiority trial to determine the capability of optical coherence tomography (OCT) imaging to show vessel morphology in comparison to imaging provided by intravascular ultrasound imaging (IVUS).

DETAILED DESCRIPTION:
Patients requiring diagnostic imaging of peripheral vessels to determine vessel condition and planning treatment strategy will have vessel segments imaged by both OCT and IVUS imaging catheters. The images will be collected into a library and independent readers will rank each image on the quality of vessel morphology and disease.

ELIGIBILITY:
Inclusion Criteria:

* adult
* suspected vascular disease that might be a candidate for IVUS
* reference vessel can accommodate imaging catheters
* successful diagnostic imaging and removal of IVUS catheter with no adverse events

Exclusion Criteria:

* if female, pregnant or breast-feeding
* unwilling to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lawson, PhD, Study Director — Avinger, Inc.
Locations (2):
- United States (2):
  - Adventis Midwest Health, Hinsdale, Illinois
  - Pottstown Hospital, Pottstown, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavillard E, Sewall L. A post-market, multi-vessel evaluation of the imaging of peripheral arteries for diagnostic purposeS comparing optical Coherence tomogrApy and iNtravascular ultrasound imaging (SCAN). BMC Med Imaging. 2020 Feb 14;20(1):18. doi: 10.1186/s12880-020-0420-7. PMID 32059702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVUS Imaging vs. OCT Imaging
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 120 matched IVUS and OCT images were collected along defined segments of peripheral vessels from 12 subjects.
Units Other Than Participants: Images
Arm/Group | IVUS Imaging vs. OCT Imaging
Number analyzed (Participants) | 12
Number analyzed (Images) | 240
Age, Continuous [Mean (Full Range); unit: years] | 68 [55 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Full Range); unit: kg] | 82 [69 to 92]
Height [Mean (Full Range); unit: cm] | 176.8 [167.6 to 187.9]
Leg of vessel accessed [Count of Participants; unit: Participants]
  Right Leg | 3
  Left Leg | 9
Vessel imaged [Number; unit: Percentage of Participants]
  SFA | 64
  Popliteal | 36
Mean length of target segment of vessel [Mean (Full Range); unit: cm] | 24 [10 to 60]
Number of images containing a specific vessel characteristic to be scored [Number; unit: Images]
  Layered Structure | 24
  Nonlayered Structure | 104
  Calcification | 40
  Stent Structure | 21
  Artifact | 120

OUTCOME MEASURES:

1. Primary Outcome: Visualization of Vessel Morphology: Layered Structure
Description: The primary endpoint was met when OCT imaging had the equivalent or lower mean score than IVUS imaging when comparing layered structures.
  Images were scored on a scale from 1 to 4. A lower score means better image quality and a higher score means worse image quality.
  Scoring Scale for image quality of layered structure:
  1. clear differentiation of vessel wall layers;
  2. differentiation of 3 wall layers;
  3. differentiation of 2 wall layers;
  4. no differentiation visible
Time Frame: During the diagnostic imaging procedures, up to 5 minutes
Population: Twenty-four imaging pairs of the 120 imaging pairs (240 images total) were analyzed for layered structures.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Images
Groups:
- IVUS Imaging: Vessel segment imaged with intravascular ultrasound (IVUS).
- OCT Imaging: Same vessel segment imaged with optical coherence tomography (OCT).
Arm/Group | IVUS Imaging | OCT Imaging
Number analyzed (Participants) | 12 | 12
Number analyzed (Images) | 24 | 24
score on a scale | 1.61 [1.48 to 1.74] | 1.49 [1.37 to 1.61]

2. Primary Outcome: Visualization of Vessel Morphology: Non-layered Structure
Description: The primary endpoint was met when OCT imaging had the equivalent or lower mean score than IVUS imaging when comparing non-layered structures.
  Images were scored on a scale from 1 to 5. A lower score means better image quality and a higher score means worse image quality.
  Scoring scale for image quality of non-layered structure:
  1-Excellent histology-like image quality to 5-unacceptably poor image quality
Time Frame: During the diagnostic imaging procedures, up to 5 minutes
Population: One hundred and four imaging pairs of the 120 imaging pairs (240 images total) were analyzed for non-layered structures.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Images
Arm/Group | IVUS Imaging | OCT Imaging
Number analyzed (Participants) | 12 | 12
Number analyzed (Images) | 104 | 104
score on a scale | 2.70 [2.53 to 2.87] | 1.82 [1.67 to 1.97]

3. Primary Outcome: Visualization of Vessel Morphology: Calcification
Description: The primary endpoint was met when OCT imaging had the equivalent or lower mean score than IVUS imaging when comparing images for calcification.
  Images were scored on a scale from 1 to 5. A lower score means better image quality and a higher score means worse image quality.
  Scoring Scale for image quality for calcification:
  1- Excellent histology-like image quality to 5- Unacceptably poor image quality.
Time Frame: During the diagnostic imaging procedures, up to 5 minutes
Population: Forty imaging pairs of the 120 imaging pairs (240 images total) were analyzed for calcification.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Images
Arm/Group | IVUS Imaging | OCT Imaging
Number analyzed (Participants) | 12 | 12
Number analyzed (Images) | 40 | 40
score on a scale | 2.45 [2.30 to 2.60] | 2.11 [1.92 to 2.30]

4. Primary Outcome: Visualization of Vessel Morphology: Stent Structure
Description: The primary endpoint was met when OCT imaging had the equivalent or lower mean score than IVUS imaging when comparing stent structure.
  Images were scored on a scale from 1 to 3. A lower score means better image quality and a higher score means worse image quality.
  Scoring Scale for image quality of Stent Structure:
  1. Excellent image;
  2. Acceptable image:
  3. Unacceptably poor image.
Time Frame: During the diagnostic imaging procedures, up to 5 minutes
Population: Twenty-one imaging pairs of the 120 imaging pairs (240 images total) were analyzed for stent structure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Images
Arm/Group | IVUS Imaging | OCT Imaging
Number analyzed (Participants) | 12 | 12
Number analyzed (Images) | 21 | 21
score on a scale | 1.79 [1.66 to 1.92] | 1.43 [1.34 to 1.55]

5. Primary Outcome: Visualization of Vessel Morphology: Artifacts
Description: The primary endpoint was met when OCT imaging had the equivalent or lower mean score than IVUS imaging when comparing imaging artifacts.
  Images were scored on a scale from 1 to 3. A lower score means better image quality and a higher score means worse image quality.
  Scoring Scale for image quality of artifacts:
  1. None;
  2. Tolerable/not limiting;
  3. Is intense and limits image quality.
Time Frame: During the diagnostic imaging procedures, up to 5 minutes
Population: One hundred and twenty imaging pairs (240 images total) were analyzed for artifacts.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Images
Arm/Group | IVUS Imaging | OCT Imaging
Number analyzed (Participants) | 12 | 12
Number analyzed (Images) | 120 | 120
score on a scale | 1.87 [1.77 to 1.97] | 1.79 [1.60 to 1.98]

6. Primary Outcome: Freedom From Adverse Events
Description: Primary safety endpoint is freedom from diagnostic imaging procedure-related and device-associated adverse events.
Time Frame: On day of diagnostic imaging procedures, up to 1 hour
Measure: Number; unit: Adverse Events
Arm/Group | IVUS Imaging | OCT Imaging
Number analyzed (Participants) | 12 | 12
Adverse Events | 0 | 0

7. Secondary Outcome: Vessel Measurement: Mean Diameter
Description: Mean diameter measurements include longest and shortest diameter at proximal, middle, and distal locations.
Time Frame: During the diagnostic imaging procedures, up to 5 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | IVUS Imaging | OCT Imaging
Number analyzed (Participants) | 12 | 12
mm
  Proximal Location: Longest Diameter | 4.7 (1.2) | 4.7 (1.0)
  Proximal Location: Shortest Diameter | 4.0 (1.1) | 3.8 (0.9)
  Middle Location: Longest Diameter | 4.3 (1.0) | 4.3 (0.9)
  Middle Location: Shortest Diameter | 3.7 (1.0) | 3.5 (0.9)
  Distal Location: Longest Diameter | 3.5 (0.9) | 3.5 (0.8)
  Distal Location: Shortest Diameter | 3.0 (0.9) | 3.1 (0.8)

8. Secondary Outcome: Vessel Measurement: Total Luminal Area
Description: Total luminal area is measured from the longest diameter at proximal, middle and distal locations.
Time Frame: During the diagnostic imaging procedures, up to 5 minutes
Measure: Mean (Standard Deviation); unit: square mm
Arm/Group | IVUS Imaging | OCT Imaging
Number analyzed (Participants) | 12 | 12
square mm
  Proximal Location: Luminal area from longest diameter | 18.55 (8.8) | 17.95 (7.3)
  Middle Location: Luminal area from longest diameter | 15.36 (6.6) | 14.83 (6.3)
  Distal Location: Luminal area from longest diameter | 10.06 (6.2) | 10.26 (5.4)

ADVERSE EVENTS:
Time Frame: On day of diagnostic imaging procedures, up to 1 hour
Description: Method of systematic assessment: any adverse events during the diagnostic imaging procedure are recorded.
Arm/Group | IVUS Imaging | OCT Imaging
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03480685/Prot_SAP_000.pdf